CLINICAL TRIAL: NCT07095816
Title: Administering Acetaminophen Orally Before Surgery Reduces Postoperative Pain in Children With Solid Tumors Under the Mode of ERAS
Brief Title: Acetaminophen Before Surgery Lowers Postop Pain in Pediatric Solid Tumor Patients (ERAS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nanjing Children's Hospital (Other)
Responsible Party: Principal Investigator, Weibing Tang, Chief of Department of neonatal surgery, Nanjing Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NCH202305012-1
Record Dates: First submitted 2025-07-13; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Analgesic; Enhanced Recovery After Surgery; Postoperative Pain; Acetaminophen; Tumor
MeSH Terms: conditions — Pain, Postoperative; Neoplasms | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acetaminophen（APAP） (Experimental): The experimental group received oral acetaminophen（10 mg/kg）two hours prior to surgery.
  Interventions: Drug: Acetaminophen
- sterilized water (Placebo Comparator): The placebo group received 10 mg/kg sterilized water two hours prior to surgery.
  Interventions: Drug: Sterilized water

INTERVENTIONS:
Drug: Acetaminophen — A prospective randomized controlled trial was conducted involving pediatric patients with solid tumors. Participants who met the inclusion criteria were randomly assigned using a computer-generated random number table. The APAP group was administered acetaminophen orally at a dose of 10 mg/kg body weight 2 hours before the surgical procedure.
  Arms: Acetaminophen（APAP）
Drug: Sterilized water — The placebo group was administered 10 mg/kg of sterile water orally two hours before the surgical procedure.
  Arms: sterilized water

SUMMARY:
Pain is the predominant subjective symptom experienced during the perioperative period in pediatric patients with solid tumors. Intense pain may impede early postoperative activities and delay the recovery process. Preemptive analgesia，as a component of multimodal analgesia strategies，aims to mitigate pain by administering analgesic interventions prior to the application of a noxious stimulus. This approach seeks to diminish both peripheral and central sensitization to pain，thereby alleviating postoperative pain. Currently，while preoperative acetaminophen is widely used in adult surgeries，research is limited for its use in pediatrics. This study aims to evaluate the impact of preemptive acetaminophen on reducing postoperative pain in children with solid tumors under the mode of ERAS.

DETAILED DESCRIPTION:
Pediatric oncology patients face unique challenges due to their distinct clinical profile. Solid tumors like neuroblastomas, teratomas, and rhabdomyosarcomas often develop in complex areas such as the retroperitoneum, pelvis, or mediastinum, where they grow invasively and can encase major blood vessels. Children typically have larger tumor-to-body size ratios than adults, necessitating more extensive surgeries and resulting in larger wounds from tumor and lymph node removal. Their poor preoperative nutrition and compromised healing abilities, due to both their disease and treatments, lead to slower wound healing and higher risk of complications.

Managing pain in pediatric cancer patients is challenging. Almost all experience pain, with over 70% facing severe pain, making it their most distressing symptom. Young children's limited cognitive abilities often lead to underreported and undertreated pain, especially after surgery. This unrelieved pain can impair breathing, hinder movement, increase infection risk, and worsen wasting. Most concerning are the potential long-term neurological effects, as significant pain in childhood may lead to lasting changes in brain structure and function.

A comprehensive meta-analysis highlights several effective preemptive analgesics, including lornoxicam, pregabalin, ibuprofen, gabapentin, and acetaminophen (APAP). APAP is particularly popular in pediatrics for its safety when properly dosed. It is quickly absorbed in the gut and metabolized in the liver, primarily by cytochrome P450 enzymes, producing a toxic intermediate, NAPQI, which is detoxified by glutathione. APAP's analgesic effects involve peripheral COX inhibition and central modulation of COX, serotonin, L-arginine/NO, endocannabinoid, and redox pathways. Preoperative APAP can prevent pain sensitization by blocking nociceptive signal transmission to the central nervous system.

APAP has proven effective for preemptive analgesia in pediatric surgeries like tonsillectomy and appendectomy, reducing pain and enhancing recovery. However, its role in pediatric oncologic surgery is unstudied, highlighting a need to explore its use in ERAS protocols for pain management in tumor resections. This study seeks to fill that gap, potentially improving perioperative pain care for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent: Written informed consent was obtained from the parents or legal guardians of all pediatric participants.

  * Age Requirement: Patients aged >1 month (infants and children) were eligible for enrollment.

    * Diagnosis & Treatment:

      * Radiologically or pathologically confirmed solid tumors. Ⅱ.Scheduled to undergo tumor resection surgery in the Department of Pediatric Surgical Oncology, Children's Hospital Affiliated to Nanjing Medical University.

Exclusion Criteria:

* Lack of Informed Consent: Parental/guardian informed consent was not obtained. ②Allergy/Intolerance: Known hypersensitivity or contraindication to acetaminophen (paracetamol).

  * Hepatic Impairment:Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels >3× the upper limit of normal (ULN).

    * Renal Dysfunction:Serum urea or creatinine levels exceeding the ULN. ⑤Recent Analgesic Use: Administration of any analgesic medication within 12 hours preoperatively.

      * PCA Exclusion: Patients not receiving postoperative intravenous patient-controlled analgesia (PCA).

Ages: 1 Month to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 182 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Using FLACC scale to assess the pain level at 1 hour after postoperative awakening | 1 hour after postoperative awakening
  The FLACC (Face, Legs, Activity, Cry, Consolability) scale score was assessed 1 hour after children aged 1 month to 6 years woke up. It evaluates five items: facial expression, leg movement, activity, crying, and consolability, each scored from 0 to 2. Total scores range from 0 to 10, with higher scores indicating greater pain: 1-3 for mild, 4-6 for moderate, and 7-10 for severe pain.
Using FLACC scale to assess the pain level at 3 hours after postoperative awakening | 3 hours after postoperative awakening
  The FLACC (Face, Legs, Activity, Cry, Consolability) scale score was assessed 3 hours after children aged 1 month to 6 years woke up. It evaluates five items: facial expression, leg movement, activity, crying, and consolability, each scored from 0 to 2. Total scores range from 0 to 10, with higher scores indicating greater pain: 1-3 for mild, 4-6 for moderate, and 7-10 for severe pain.
Using FLACC scale to assess the pain level at 6 hours after postoperative awakening | 6 hours after postoperative awakening
  The FLACC (Face, Legs, Activity, Cry, Consolability) scale score was assessed 6 hours after children aged 1 month to 6 years woke up. It evaluates five items: facial expression, leg movement, activity, crying, and consolability, each scored from 0 to 2. Total scores range from 0 to 10, with higher scores indicating greater pain: 1-3 for mild, 4-6 for moderate, and 7-10 for severe pain.
Using FLACC scale to assess the pain level at 12 hours after postoperative awakening | 12 hours after postoperative awakening
  The FLACC (Face, Legs, Activity, Cry, Consolability) scale score was assessed 12 hours after children aged 1 month to 6 years woke up. It evaluates five items: facial expression, leg movement, activity, crying, and consolability, each scored from 0 to 2. Total scores range from 0 to 10, with higher scores indicating greater pain: 1-3 for mild, 4-6 for moderate, and 7-10 for severe pain.
Using FLACC scale to assess the pain level at 24 hours after postoperative awakening | 24 hours after postoperative awakening
  The FLACC (Face, Legs, Activity, Cry, Consolability) scale score was assessed 24 hours after children aged 1 month to 6 years woke up. It evaluates five items: facial expression, leg movement, activity, crying, and consolability, each scored from 0 to 2. Total scores range from 0 to 10, with higher scores indicating greater pain: 1-3 for mild, 4-6 for moderate, and 7-10 for severe pain.
Using FLACC scale to assess the pain level at 48 hours after postoperative awakening | 48 hours after postoperative awakening
  The FLACC (Face, Legs, Activity, Cry, Consolability) scale score was assessed 48 hours after children aged 1 month to 6 years woke up. It evaluates five items: facial expression, leg movement, activity, crying, and consolability, each scored from 0 to 2. Total scores range from 0 to 10, with higher scores indicating greater pain: 1-3 for mild, 4-6 for moderate, and 7-10 for severe pain.
Using NRS scale to assess the pain level at 1 hour after postoperative awakening | 1 hour after postoperative awakening
  The NRS (Numerical Rating Scale) pain score was assessed 1 hour after children aged 6 years and above woke up. Total scores range from 0 (no pain) to 10 (most severe pain). Scores are categorized as 1-3 for mild, 4-6 for moderate, and 7-10 for severe pain.
Using NRS scale to assess the pain level at 3 hours after postoperative awakening | 3 hours after postoperative awakening
  The NRS (Numerical Rating Scale) pain score was assessed 3 hours after children aged 6 years and above woke up. Total scores range from 0 (no pain) to 10 (most severe pain). Scores are categorized as 1-3 for mild, 4-6 for moderate, and 7-10 for severe pain.
Using NRS scale to assess the pain level at 6 hours after postoperative awakening | 6 hours after postoperative awakening
  The NRS (Numerical Rating Scale) pain score was assessed 6 hours after children aged 6 years and above woke up. Total scores range from 0 (no pain) to 10 (most severe pain). Scores are categorized as 1-3 for mild, 4-6 for moderate, and 7-10 for severe pain.
Using NRS scale to assess the pain level at 12 hours after postoperative awakening | 12 hours after postoperative awakening
  The NRS (Numerical Rating Scale) pain score was assessed 12 hours after children aged 6 years and above woke up. Total scores range from 0 (no pain) to 10 (most severe pain). Scores are categorized as 1-3 for mild, 4-6 for moderate, and 7-10 for severe pain.
Using NRS scale to assess the pain level at 24 hours after postoperative awakening | 24 hours after postoperative awakening
  The NRS (Numerical Rating Scale) pain score was assessed 24 hours after children aged 6 years and above woke up. Total scores range from 0 (no pain) to 10 (most severe pain). Scores are categorized as 1-3 for mild, 4-6 for moderate, and 7-10 for severe pain.
Using NRS scale to assess the pain level at 48 hours after postoperative awakening | 48 hours after postoperative awakening
  The NRS (Numerical Rating Scale) pain score was assessed 48 hours after children aged 6 years and above woke up. Total scores range from 0 (no pain) to 10 (most severe pain). Scores are categorized as 1-3 for mild, 4-6 for moderate, and 7-10 for severe pain.

SECONDARY OUTCOMES:
The number of patient-controlled analgesia (PCA) pump activations | during the first 48 postoperative hours
  The number of patient-controlled analgesia (PCA) pump activations within 48 hours postoperatively
Serum Alanine Aminotransferase (ALT) Concentration | 24 hours after surgery
  alanine aminotransferase
Serum Aspartate Aminotransferase (AST) Concentration | 24 hours after surgery
  aspartate aminotransferase
Serum Urea Concentration | 24 hours after surgery
  urea
Plasma Creatinine Concentration | 24 hours after surgery
  creatinine values
Serum Procalcitonin Concentration (ng/mL) | 24 hours after surgery
  Postoperative inflammatory markers including procalcitonin, C-reactive protein, white blood cell count, absolute neutrophil count, absolute lymphocyte count, and neutrophil-to-lymphocyte ratio.
Serum C-Reactive Protein Concentration (mg/L) | 24 hours after surgery
  Postoperative inflammatory markers including procalcitonin, C-reactive protein, white blood cell count, absolute neutrophil count, absolute lymphocyte count, and neutrophil-to-lymphocyte ratio.
Peripheral White Blood Cell Count (×10⁹/L) | 24 hours after surgery
  Postoperative inflammatory markers including procalcitonin, C-reactive protein, white blood cell count, absolute neutrophil count, absolute lymphocyte count, and neutrophil-to-lymphocyte ratio.
Absolute Neutrophil Count (×10⁹/L) | 24 hours after surgery
  Postoperative inflammatory markers including procalcitonin, C-reactive protein, white blood cell count, absolute neutrophil count, absolute lymphocyte count, and neutrophil-to-lymphocyte ratio.
Absolute Lymphocyte Count (×10⁹/L) | 24 hours after surgery
  Postoperative inflammatory markers including procalcitonin, C-reactive protein, white blood cell count, absolute neutrophil count, absolute lymphocyte count, and neutrophil-to-lymphocyte ratio.
Neutrophil-to-Lymphocyte Ratio | 24 hours after surgery
  Postoperative inflammatory markers including procalcitonin, C-reactive protein, white blood cell count, absolute neutrophil count, absolute lymphocyte count, and neutrophil-to-lymphocyte ratio.
Intraoperative Respiratory Rate (breaths per minute) | during the operation
  Intraoperative monitoring of respiratory rate, heart rate, systolic blood pressure, and diastolic blood pressure was performed in pediatric patients throughout the surgical procedure.
Intraoperative Heart Rate (beats per minute) | during the operation
  Intraoperative monitoring of respiratory rate, heart rate, systolic blood pressure, and diastolic blood pressure was performed in pediatric patients throughout the surgical procedure.
Intraoperative Systolic Blood Pressure (mmHg) | during the operation
  Intraoperative monitoring of respiratory rate, heart rate, systolic blood pressure, and diastolic blood pressure was performed in pediatric patients throughout the surgical procedure.
Intraoperative Diastolic Blood Pressure (mmHg) | during the operation
  Intraoperative monitoring of respiratory rate, heart rate, systolic blood pressure, and diastolic blood pressure was performed in pediatric patients throughout the surgical procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Weibing Tang, Study Chair — Children's Hospital of Nanjing Medical University
Locations (1):
- Children's Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (including demographic, clinical, and outcome variables) collected during the trial will be made available to qualified researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become accessible:Starting Date: 6 months after study completion；End Date: Minimum 5 years after publication
Access Criteria: Access to IPD requires submitting a formal research proposal (including hypothesis/analysis plan, ethical approval proof if applicable, and conflict of interest disclosure) to the investigator's email, along with a signed Data Use Agreement (DUA) prohibiting re-identification, commercial use, and redistribution.